CLINICAL TRIAL: NCT00899457
Title: Molecular Predictors of Lung Cancer Behavior: Controls
Brief Title: Molecular Markers in Predicting Lung Cancer Development Using Tissue Samples From Healthy Participants
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pierre P. Massion, MD, Associate Professor of Medicine (Allergy, Pulmonary & Critical Care) and Cancer Biology; Pulmonary and Critical Care Medicine Doctor, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 0734; P50CA090949 (NIH); P30CA068485 (NIH); VU-VICC-THO-0734; VICC-THO-0734
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2013-04

CONDITIONS: Healthy, no Evidence of Disease; Lung Cancer
Keywords: squamous cell lung cancer; non-small cell lung cancer; small cell lung cancer; healthy, no evidence of disease
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy, non-smokers
  Interventions: Genetic: proteomic profiling; Other: biologic sample preservation procedure; Other: laboratory biomarker analysis; Procedure: bronchoscopy

INTERVENTIONS:
Genetic: proteomic profiling — Collection of tissue, blood, urine, mouth cells, spit, nasal airway cells and breath
Other: biologic sample preservation procedure — Collection of tissue, blood, urine, mouth cells, spit, nasal airway cells and breath
Other: laboratory biomarker analysis — Collection of tissue, blood, urine, mouth cells, spit, nasal airway cells and breath
Procedure: bronchoscopy — Collection of breath condensate.

SUMMARY:
RATIONALE: Studying samples of blood, urine, sputum, mouth cells, and bronchial tissue from healthy participants in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors learn more about the development of cancer.

PURPOSE: This laboratory study is looking for molecular markers in predicting lung cancer development using tissue samples from healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain biological specimens from healthy participants with no known risk of lung cancer to use as controls in the study of lung cancer progression.
* To identify new molecular abnormalities specific to the development of squamous cell carcinoma of the lung.

OUTLINE: Serum, urine, sputum, and buccal cell samples are collected. Patients also undergo bronchoscopy for collection of bronchial tissue and bronchial brush samples. The samples are used for genomic and proteomic studies to identify new molecular abnormalities specific to the development of lung cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participant

  * No history of smoking
  * No history of cancer

PATIENT CHARACTERISTICS:

* SWOG performance status 0
* No clinically apparent bleeding diathesis

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, non-smokers.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Collection of biological specimens to use as controls in the study of lung cancer progression | Off study date, up to one year
  Specimens are collected from healthy participants with no known risk of lung cancer

SECONDARY OUTCOMES:
Identification of new molecular abnormalities specific to the development of squamous cell carcinoma of the lung | off-study date, up to one year
Selection of important genes/proteins differentially expressed between study groups (e.g., normal vs low-grade vs high-grade vs invasive) and between normal smokers vs normal non-smokers | off-study date, up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre P. Massion, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee